CLINICAL TRIAL: NCT01936337
Title: A Multi-center, Double-blinded, Randomized, Placebo-controlled, Phase II Study to Evaluate the Safety, Tolerability and Efficacy of a Topical Application of DLX105 Onto Lesional Skin in Patients With Mild-to-moderate Psoriasis Vulgaris
Brief Title: Topical Double-blind, Randomized, Placebo-controlled Study in Psoriasis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Delenex Therapeutics AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DLX105-003-002-001
Record Dates: First submitted 2013-08-28; First posted 2013-09-06 (Estimated); Last update posted 2014-08-12 (Estimated); Status verified 2014-08

CONDITIONS: Psoriasis Vulgaris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DLX105 Hydrogel (Active Comparator)
  Interventions: Drug: DLX105 Hydrogel
- Placebo Hydrogel (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DLX105 Hydrogel — topical administration on psoriatic plaque
  Arms: DLX105 Hydrogel
Drug: Placebo — topical administration on psoriatic plaque
  Arms: Placebo Hydrogel

SUMMARY:
In this study, the safety, tolerability and efficacy of DLX105 administered topically onto the psoriatic lesion of mild-to-moderate psoriasis patients will be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent prior to initiation of any study procedures.
2. Male or female Caucasian aged 18-75 years.
3. Male or female patients with stable chronic mild-to-moderate plaque-type psoriasis (PASI ≤15).
4. Male or female Caucasian patients with stable chronic mild-to-moderate plaque-type psoriasis (PASI ≤15) aged 18-75 years who must have at least two psoriasis lesions of >9 cm2 (located at arms and/or trunk, excluding elbows and legs), stable for at least 3 months, local PASI score ≥8.
5. Affected body surface area (BSA) ≤10%.
6. Negative pregnancy test for females of child-bearing potential (pre-menopausal, <2 years post-menopausal, not surgically sterile).
7. Willing and able to participate in the trial as an outpatient and comply with all trial requirements.

Exclusion Criteria:

1. Forms of psoriasis other than chronic plaque-type only (e.g., pustular, erythrodermic and guttate psoriasis, palmar, plantar or nail disease) at screening.
2. Drug-induced psoriasis (i.e., new onset or current exacerbation from beta-blockers, calcium channel inhibitors or lithium) prior to randomization
3. Ongoing use of prohibited psoriasis treatments (duration of washout, i.e. discontinuation prior to randomization):

   1. Biological agents, e.g. adalimumab, etanercept, infliximab, ustekinumab, alefacept (12 weeks)
   2. Systemic therapy for psoriasis and psoriatic arthritis (other than above) e.g. methotrexate, cyclosporin, fumaric acid (derivatives), systemic steroids (4 weeks)
   3. Photochemotherapy e.g., ultraviolet A with psoralen (PUVA) (4 weeks)
   4. Phototherapy e.g., ultraviolet A (UVA) or ultraviolet B (UVB) (2 weeks)
   5. Topical therapies for the treatment of Ps such as corticosteroids, vitamin D analogues or retinoids within 14 days prior to baseline
   6. Other investigational psoriasis drugs (4 weeks or 5 half-lives, whichever is longer)
4. Intake of any investigational drug or participation in a Clinical Trial within 4 weeks or 5 half-lives, (whichever is longer) prior to baseline.
5. History or evidence of active tuberculosis. All patients will be tested for tuberculosis status using a blood test (QuantiFERON TB-Gold) unless this test has been performed within 4 months prior to randomization and was negative. Patients with evidence of latent tuberculosis may enter the trial after sufficient treatment has been initiated according to local regulations.
6. Active systemic infections (other than common cold) during the two weeks before randomization
7. Positive test for hepatitis B or C at screening
8. Positive test for HIV at screening
9. History or symptoms of malignancy of any organ system (other than history of basal cell carcinoma and / or up to three squamous cell carcinomas of the skin, if successful treatment has been performed, with no signs of recurrence; actinic keratosis, if present at screening, should be treated according to standard therapy before randomization), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
10. History of severe hypersensitivity to any human or humanized biological agents
11. Any severe, progressive or uncontrolled medical condition at baseline that in the judgment of the investigator prevents the patient from participating in the study.
12. Any clinically significant abnormal laboratory tests at screening
13. Active liver disease with alanine aminotransferase (ALT) and / or aspartate aminotransferase (AST) > 3 x upper limit of normal at screening
14. History of moderate or severe congestive heart failure (New York Heart Association [NYHA] class III or IV)
15. Inability or unwillingness to undergo repeated venipunctures (e.g., due to poor tolerability or lack of access to veins)
16. History or evidence of drug or alcohol abuse within the 6 months prior first study drug administration
17. Patients who had live vaccination within 6 weeks prior first study drug administration, or will require live vaccination during the course of the trial
18. History of hypersensitivity to any of the excipients of the study drugs or to excipients of similar chemical classes
19. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (HCG) laboratory test (> 5 mIU/mL)
20. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant. UNLESS they are women whose partners have been sterilized by vasectomy

    1. Using a highly effective method of birth control (i.e. one that results in a less than 1% per year failure rate when used consistently and correctly, such as implants, injectables, combined oral contraceptives, condoms (by the partner), and intrauterine devices (IUDs)). Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not considered acceptable forms of birth control within this study
    2. Reliable contraception should be maintained throughout the study and for 2 weeks after the last study drug administration

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2013-08; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Assessment of local tolerability by the investigator | up to 6 weeks
  using a validated score for each treatment area
assessment of local tolerability sensations by the patient | up to 6 weeks
  using a visual analogue scale for each treatment area
collection of Adverse Events | up to 6 weeks
Determination of efficacy of DLX105 as compared to baseline | Baseline to Week 4
  assessment of Local PASI score per plaque measured at week 4 compared to baseline
Determination of efficacy of DLX105 as compared to Placebo at week 4 | baseline to week 4
  Local PASI difference at week 4 between DLX105 and placebo

SECONDARY OUTCOMES:
Detection of Immunogenicity | up to 6 weeks
  Anti-drug-antibodies will be determined to assess the immunogenic potential of DLX105.
Detection of Pharmacokinetics | up to 6 weeks
  Pharmacokinetics through levels will be measured in serum at 4 time points over 6 weeks.

CONTACTS AND LOCATIONS:
Locations (3):
- University Hospital AKH, Vienna, Austria
- Germany (2):
  - University Hospital, Münster
  - University Hospital, Tübingen